CLINICAL TRIAL: NCT04172961
Title: A Phase 4 Study to Assess the Clinical Efficacy of Nanomicellular Cyclosporine 0.09% Versus Lifitegrast 5.0% for Central Corneal Stain Clearing Over 90 Days
Brief Title: Clinical Efficacy of Two Topical Dry Eye Drops for Central Corneal Stain Clearing Over 90 Days
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toyos Clinic (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUNTC-001
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins; lifitegrast

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: study medication will be provided in an unmarked box with tape externally covering any identifying language
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nanomicellular Cyclosporine 0.09 prior to surgery (Experimental): 50 subjects receive nanomicellular cyclosporien 0.09% prior to elective ophthalmic surgery
  Interventions: Drug: nanomicellular cyclosporine 0.09%
- Lifitegrast 5.0% (Active Comparator): 50 subjects receive liftigrast 5.0% prior to elective ophthalmic surgery
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: nanomicellular cyclosporine 0.09% — topical ophthalmic drop prior to elective surgery for eligible patients
  Other Names: Cequa
  Arms: Nanomicellular Cyclosporine 0.09 prior to surgery
Drug: Lifitegrast — topical ophthalmic drop prior to elective surgery for eligible patients
  Other Names: Xiidra
  Arms: Lifitegrast 5.0%

SUMMARY:
This study will be a randomized, double-blind prospective in 3 clinical sites to compare the efficacy of two currently approved topical ophthalmic drops in the clearing central corneal staining in 90 days prior to elective cataract or LASIK surgery.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind prospective study in 3 sites in the US to compare efficacy of improvement in central corneal staining with fluorescein dye evaluations at slit lamp exam, secondarily improvement in OSDI questionnaire with additional questions regarding dysgeusia, blurriness, and sensation of burning, improvements in corneal topography and improvements in Schirmer's testing. 100 study subjects 18-85 male or female will be enrolled in the Nashville, Beverly Hills and St. Louis areas who are generally healthy with central corneal staining and scheduled for uncomplicated phacoemulsification or uncomplicated LASIK.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read, understand and sign informed consent.
2. Provision of signed and dated informed consent and HIPAA authorization .
3. Willingness to comply with study procedures and availabilty for duration of study.
4. Aged 18-85, male or female
5. Minimum of 5 central corneal superficial punctate keratitis spots.
6. Normal eyelid anatomy
7. highly effective contraception for at least 1 month prior to screening and agreement to use effective contraception during study participation and for an additional 4 weeks after study drug discontinuation.
8. Postmenopausal or surgical sterilization.

   -

Exclusion Criteria:

1. Known hypersensitivity or contraindication to investigational product.
2. Contact lens use within one month prior to screening
3. Unwilling to discontinue contact lens.
4. pregnancy or lactation.
5. topical or nasal vasoconstrictors within 14 days prior to screening or unable to refrain from same.
6. Ocular surgery or eyelid surgery within 6 months prior to screening
7. Subjects can be on the following medications if they have been on a stable dose for 12 weeks: loteprednol, tetracycline, omega 3, anticholinergics, anticonvulsants, antidepressants, retinoids, systemic immunosuppressives including oral steroids, non-steroidals, antihistamines, mast cell stabilizers, punctal plugs, corticotropin repository or glaucoma medications.
8. abstain from eyelast growth products containing prostaglandin
9. Must not have had penetrating intraocular surgery, refractive surgery, cornea transplant, eyelid surgery within 6 months prior to Visit 1
10. Febrile illness within 1 week
11. Treatment with another investigational drug or intervention within one month
12. History of herpetic keratitis.
13. Serious or severe disease or uncontrolled medical condition that in the judgment of the investigator could confound study study assessments or limit compliance.
14. Use of new prescription eyedrop within 90 days of screening.
15. Change in systemic medication within 90 days of screening
16. Anticipated relocation or extensive travel during study period. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
change in central corneal staining | 90 days
  use of fluorescein staining to count at slit lamp actual number of central cornea spk

SECONDARY OUTCOMES:
change in OSDI questionnaire with additional questions of dysgeusia, blurriness and sensation of burning | 90 days
  subjective improvement of symptoms and assessment of adverse events
change in corneal topography | 90 days
  variation in measurements of corneal topography
change in Schirmers testing | 90 days
  change in Schirmers testing

CONTACTS AND LOCATIONS:
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual date with other researchers